CLINICAL TRIAL: NCT04687540
Title: Meal-regulated Substrate Metabolism, Influence of Obesity and IL-6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Helga Ellingsgaard, Group leader, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: METO
Record Dates: First submitted 2020-12-17; First posted 2020-12-29 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Obesity; Healthy
Keywords: Interleukin-6; Tocilizumab; Postprandial; Postabsorptive; Substrate metabolism; Fat metabolism; Glucose metabolism; Protein metabolism; Isotope dilution technique
MeSH Terms: conditions — Obesity | interventions — tocilizumab; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study is designed in a placebo-controlled crossover manner, consisting of a screening visit and two study visits. Due to the 4-week wash out period of the IL-6 receptor antibody tocilizumab, the order of study visits will be identical in all subjects; hence, study visits will not be randomized. Subjects will be infused with tocilizumab at the end of study visit 1. This will allow us to study the effect of tocilizumab on study visit 2.
Who Masked: Participant
Masking Description: Only subjects will be masked regarding order of saline and tocilizumab infusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study day 1 (study visit 1) (Placebo Comparator): Baseline measurements (pre-intervention) are obtained on study visit 1.
  Interventions: Drug: Tocilizumab
- Study day 21 (study visit 2) (Active Comparator): Post-intervention measurements: Participants will be under the influence of tocilizumab, which was injected at the end of study visit 1.
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Tocilizumab — Baseline: Tocilizumab (infusion of 8 mg/kg bodyweight or a maximum of 800 mg) will be infused over 60 minutes at the end for the study day, therefore study visit 1 (study day 1) measurements are baseline.
  Other Names: RoActemra
  Arms: Study day 1 (study visit 1)
Drug: Saline 0.9% — Participants are under influence of tocilizumab since the effect of the drug will last for 4 weeks. Participants will be infused with saline at study visit 2 (study day 21). Placebo to tocilizumab will be saline (NaCl 0.9%) as tocilizumab is a colorless solution and has to be diluted with NaCl 0.9% prior to administration
  Arms: Study day 21 (study visit 2)

SUMMARY:
The overall purpose of this explorative yet quantitative study project is to understand how blocking IL-6 signaling leads to the expansion of adipose tissue mass in humans in vivo. The aim is to gain in depth knowledge about how IL-6 receptor blockade affects human lipid, glucose and protein metabolism, specifically the uptake and storage of substrates from a meal vs. their utilization, hence the balance determining whether one gains or loses fat mass.

DETAILED DESCRIPTION:
Lacking IL-6 signaling leads to an expansion of adipose tissue mass in rodents and humans. However, the underlying mechanisms have not been identified.This project aims to investigate the overall hypothesis that IL-6 receptor blockade changes substrate metabolism during postabsorptive and postprandial states to favor storage over mobilization of fat and to favor glucose over fat as a source for energy production. This hypothesis finds some support in the literature: Infusion of recombinant IL-6 into humans, leading to high concentrations of IL-6 in the circulation, stimulates lipolysis and free fatty acid oxidation.

Therefore, the investigators hypothesize that IL-6 receptor blockade impairs the mobilization of FFA from adipose tissue and impairs fat oxidation in skeletal muscle in the postabsorptive state. In the postprandial, state the investigators hypothesize that IL-6 receptor blockade reduces the insulin-induced uptake and deposition of fat by adipose tissue and skeletal muscle, therefore contributing to ectopic fat deposition in the liver.

In this study 12 lean and 12 obese male participants will be included. The participants will attend one screening visit and two study visits. The IL-6 receptor antibody tocilizumab will be infused on study visit 1.

Isotope dilution techniques, blood flow measurements, arterio-venous differences across adipose tissue and skeletal muscle, fat and skeletal muscle biopsies will be used to assess lipid, glucose and protein kinetics on a whole-body as well as fat and skeletal muscle level in the fasting state and after the ingestion of a liquid mixed-meal. Respiratory exchange ratio will be measured by indirect calorimetry.

ELIGIBILITY:
Inclusion Criteria:

Healthy males:

* Age ≥ 18 years and ≤ 40 years
* BMI < 18 and > 25 kg/m2
* Healthy (based on screening)
* Stable body weight for 6 months

Obese males:

* Age ≥ 18 years and ≤ 40 years
* BMI ≥ 30 and ≤ 40 kg/m2
* Healthy (based on screening)
* Stable body weight for 6 months

Exclusion Criteria:

* Smoking
* Evidence of severe thyroid or heart disease, inflammatory diseases, current infection, liver disease (transaminases >2x upper normal range), kidney disease (creatinine >1.5 mg/dl), known immunosuppressive disease, corticosteroid use, regular NSAID or paracetamol usage, aspirin use >100 mg/d, history of carcinoma, history of tuberculosis, anemia (hematocrit <33%), WBC <2 x 10^3/ul, platelets <100 x 10^3/ul, bleeding disorders, obstructive pulmonary disease
* Femoral hernia, vascular prosthesis, vascular thrombosis
* Previous nerve damage, many previous femoral catheter installations

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Whole-body, fat and skeletal muscle fat turnover | 0-21 days
  Rate of appearance and disappearance of glycerol and palmitate, fatty acid oxidation and re-esterification, arterio-venous differences of glycerol, palmitate, triglycerides across adipose tissue and skeletal muscle, triglycerides fractional synthesis rate in the postabsorptive and postprandial state in the presence of tocilizumab as compared to placebo
Whole-body, fat and skeletal muscle glucose turnover | 0-21 days
  Rate of appearance and disappearance of glucose, arterio-venous differences of glucose across adipose tissue and skeletal muscle, glycogen fractional synthesis rate in the postabsorptive and postprandial state in the presence of tocilizumab as compared to placebo
Whole-body, fat and skeletal muscle amino acid and protein turnover | 0-21 days
  Rate of appearance and disappearance of amino acids, arterio-venous differences of amino acids across adipose tissue and skeletal muscle, protein fractional synthesis rate in the postabsorptive and postprandial state, in the presence of tocilizumab as compared to placebo
Nutrient uptake | 0-21 days
  Uptake of fatty acids, glucose and amino acids from a meal in the presence of tocilizumab as compared to placebo

SECONDARY OUTCOMES:
Free fatty acids (FFA) (plasma concentration) | 0-21 days
  Change in postabsorptive and postprandial FFA levels in the presence of tocilizumab as compared to placebo
Triglycerides (plasma concentration) | 0-21 days
  Change in postabsorptive and postprandial triglycerides levels in the presence of tocilizumab as compared to placebo
Subjective feeling of hunger and fullness | 0-21 days
  Hunger and fullness will be assessed on a VAS scale.
Insulin (plasma concentration) | 0-21 days
  Change in postabsorptive and postprandial insulin levels in the presence of tocilizumab as compared to placebo
C-peptide (plasma concentration) | 0-21 days
  Change in postabsorptive and postprandial c-peptide levels in the presence of tocilizumab as compared to placebo
Glucagon (plasma concentration) | 0-21 days
  Change in postabsorptive and postprandial glucagon levels in the presence of tocilizumab as compared to placebo
Cortisol (plasma concentration) | 0-21 days
  Change in postabsorptive and postprandial cortisol levels in the presence of tocilizumab as compared to placebo
Adrenaline (plasma concentration) | 0-21 days
  Change in postabsorptive and postprandial adrenaline levels in the presence of tocilizumab as compared to placebo
Noradrenaline (plasma concentration) | 0-21 days
  Change in postabsorptive and postprandial noradrenaline levels in the presence of tocilizumab as compared to placebo
Cytokines, incl. interleukin-6 (IL-6) (plasma concentration) | 0-21 days
  Change in postabsorptive and postprandial cytokine levels in the presence of tocilizumab as compared to placebo
Total and active GLP-1 (plasma concentration) | 0-21 days
  Change in postabsorptive and postprandial total and active GLP-1 levels in the presence of tocilizumab as compared to placebo
GIP (plasma concentration) | 0-21 days
  Change in postabsorptive and postprandial GIP levels in the presence of tocilizumab as compared to placebo
PYY (plasma concentration) | 0-21 days
  Change in postabsorptive and postprandial PYY postabsorptive and postprandial in the presence of tocilizumab as compared to placebo
Leptin (plasma concentration) | 0-21 days
  Change in postabsorptive and postprandial leptin levels in the presence of tocilizumab as compared to placebo
Testosterone (plasma concentration) | 0-21 days
  Change in postabsorptive testosterone levels in the presence of tocilizumab as compared to placebo
TSH (plasma concentration) | 0-21 days
  Change in postabsorptive TSH levels in the presence of tocilizumab as compared to placebo
GH (plasma concentration) | 0-21 days
  Change in postabsorptive and postprandial GH levels in the presence of tocilizumab as compared to placebo
Respiratory exchange ratio (RER) | 0-21 days
  Indirect calorimetry measured in post-absorptive and postprandial states
Femoral artery blood flow | 0-21 days
  Change in femoral artery blood flow in the presence of tocilizumab as compared to placebo
RNA sequencing | 0-21 days
  RNA sequencing on adipose tissue and skeletal muscle biopsies, monocytes with or without the influence of tocilizumab
Mitochondrial respiration (Oroboros) | 0-21 days
  Mitochondrial respiration in skeletal muscle biopsies with or without the influence of tocilizumab
Gastric emptying rate | 0-21 days
  Gastric emptying rate in the presence of tocilizumab as compared to placebo
Plasma metabolome | 0-21 days
  Plasma metabolome with or without the influence of tocilizumab
Plasma, lipidome | 0-21 days
  Plasma lipidome with or without the influence of tocilizumab
Adipose tissue proteome | 0-21 days
  Adipose tissue proteome with or without the influence of tocilizumab
Skeletal muscle proteome | 0-21 days
  Skeletal muscle proteome with or without the influence of tocilizumab
Monocyte secretome | 0-21 days
  Change in the postabsorptive and postprandial secretory profile of monocytes in the presence of tocilizumab as compared to placebo
IL-6 signaling activation in monocytes | 0 days
  IL-6 signaling pathway activation in monocytes from lean participants compared to from obese participants

CONTACTS AND LOCATIONS:
Overall Officials: Helga Ellingsgaard, PhD, Principal Investigator — CFAS, Rigshospitalet
Locations (1):
- Rigshospitalet, Centre of Inflammation and Metabolism (CIM) Centre for Physical Activity Research (CFAS), Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wallenius V, Wallenius K, Ahren B, Rudling M, Carlsten H, Dickson SL, Ohlsson C, Jansson JO. Interleukin-6-deficient mice develop mature-onset obesity. Nat Med. 2002 Jan;8(1):75-9. doi: 10.1038/nm0102-75. PMID 11786910
- [Background] Wueest S, Item F, Boyle CN, Jirkof P, Cesarovic N, Ellingsgaard H, Boni-Schnetzler M, Timper K, Arras M, Donath MY, Lutz TA, Schoenle EJ, Konrad D. Interleukin-6 contributes to early fasting-induced free fatty acid mobilization in mice. Am J Physiol Regul Integr Comp Physiol. 2014 Jun 1;306(11):R861-7. doi: 10.1152/ajpregu.00533.2013. Epub 2014 Apr 2. PMID 24694381
- [Background] Wedell-Neergaard AS, Lang Lehrskov L, Christensen RH, Legaard GE, Dorph E, Larsen MK, Launbo N, Fagerlind SR, Seide SK, Nymand S, Ball M, Vinum N, Dahl CN, Henneberg M, Ried-Larsen M, Nybing JD, Christensen R, Rosenmeier JB, Karstoft K, Pedersen BK, Ellingsgaard H, Krogh-Madsen R. Exercise-Induced Changes in Visceral Adipose Tissue Mass Are Regulated by IL-6 Signaling: A Randomized Controlled Trial. Cell Metab. 2019 Apr 2;29(4):844-855.e3. doi: 10.1016/j.cmet.2018.12.007. Epub 2018 Dec 27. PMID 30595477
- [Background] Christensen RH, Lehrskov LL, Wedell-Neergaard AS, Legaard GE, Ried-Larsen M, Karstoft K, Krogh-Madsen R, Pedersen BK, Ellingsgaard H, Rosenmeier JB. Aerobic Exercise Induces Cardiac Fat Loss and Alters Cardiac Muscle Mass Through an Interleukin-6 Receptor-Dependent Mechanism: Cardiac Analysis of a Double-Blind Randomized Controlled Clinical Trial in Abdominally Obese Humans. Circulation. 2019 Nov 12;140(20):1684-1686. doi: 10.1161/CIRCULATIONAHA.119.042287. Epub 2019 Nov 11. No abstract available. PMID 31710522
- [Background] Petersen EW, Carey AL, Sacchetti M, Steinberg GR, Macaulay SL, Febbraio MA, Pedersen BK. Acute IL-6 treatment increases fatty acid turnover in elderly humans in vivo and in tissue culture in vitro. Am J Physiol Endocrinol Metab. 2005 Jan;288(1):E155-62. doi: 10.1152/ajpendo.00257.2004. Epub 2004 Sep 21. PMID 15383370
- [Background] van Hall G, Steensberg A, Sacchetti M, Fischer C, Keller C, Schjerling P, Hiscock N, Moller K, Saltin B, Febbraio MA, Pedersen BK. Interleukin-6 stimulates lipolysis and fat oxidation in humans. J Clin Endocrinol Metab. 2003 Jul;88(7):3005-10. doi: 10.1210/jc.2002-021687. PMID 12843134
- [Derived] Trinh B, Rasmussen SJ, Brogger-Jensen ME, Engelhard CA, Lund A, Tavanez AR, Vassilieva A, Janum S, Iepsen UW, Kiens B, Moller K, Pedersen BK, Van Hall G, Ellingsgaard H. Inhibition of basal IL-6 activity promotes subcutaneous fat retention in humans during fasting and postprandial states. Cell Rep Med. 2025 Apr 15;6(4):102042. doi: 10.1016/j.xcrm.2025.102042. Epub 2025 Mar 26. PMID 40147447